CLINICAL TRIAL: NCT06772987
Title: Safety and Efficacy of an Accelerated, Rectangular Waveform rTMS Protocol in Treatment of Adults With Major Depressive Disorder
Brief Title: NQ TMS for MDD Therapy Using 1 Day x 3 Sessions Protocol for Adult Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeuroQore Inc. (Industry)
Collaborators: Makromed Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-NQ-2024-01; BRANY IRB File #24-02-624-1959 (Other: Biomedical Research Alliance of New York (BRANY))
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Major Depressive Disorder; Accelerated Treatment; 1-Day Treatment
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Accelerated Protocol (Experimental): 1 Day x 3 Sessions treatment protocol, with 60 minutes rest between sessions. Each session is a 19-minutes rTMS treatment.
  Interventions: Device: Accelerated rTMS treatment

INTERVENTIONS:
Device: Accelerated rTMS treatment — 1 Day x 3 Sessions of 19-minutes rTMS treatment, with 60 minutes rest between sessions.

SUMMARY:
Transcranial Magnetic Stimulation (TMS) Therapy is a non-invasive procedure that uses magnetic pulses to stimulate the cortex (brain) to treat Major Depressive Disorder (MDD). Currently established therapy uses one 19-minute treatment session per day for 5 days per week for 6 weeks, for a total of 30 treatment sessions.

The goal of this clinical trial is to evaluate the safety and effectiveness of an accelerated but shortened TMS dosing regimen for adults with MDD aged 22-85.

Participants in this study will be subjected to the same 19-minutes treatment session, but three times on the same day, and only for one day. This will greatly reduce the logistical burden of completing the therapy regime.

DETAILED DESCRIPTION:
Study Description:

This single center, open label study will evaluate the safety and efficacy of accelerating the delivery of the NeuroQore TMS system's rectangular waveform rTMS protocol for the treatment of adults with MDD aged 22-85.

Currently cleared protocol with the FDA (the Standard of Care Protocol) is one 19-min treatment session a day for 5 days/week for 6 weeks. The accelerated protocol will involve the same 19-min treatment session offered three times in a single day, with no additional treatment sessions.

Primary Objectives:

1. To assess the efficacy of the NeuroQore TMS system, with accelerated delivery in the treatment of adults with MDD, as measured by a change in MADRS score 24 hours and 7 days after the treatment end.
2. To compare the safety profile of the accelerated delivery protocol to the historical safety profile of the Standard of Care protocol.

Endpoints:

Primary

* Change in MADRS score from baseline to 24 hours and 7 days post-treatment.
* Number and type of adverse events. Secondary
* Change in PHQ-9 score from baseline to 24 hours and 7 days post-treatment.

Study Population:

Men and women 22-85 with MDD that have failed one medication in the current episode.

Study Intervention:

NeuroQore TMS System includes (1) a pulse generator, (2) a magnetic coil, (3) a coil cooler, and (4) a chair with a headpiece. It has been cleared for clinical use (K232688) by the FDA for the treatment of MDD using a 19-min Standard of Care protocol.

Treatment during this study will be administered according to this protocol and following the instructions in the device user manual. Personalized stimulation targets will be produced from participants' structural MRI via the proprietary targeting generation component of the NeuroQore TMS system.

Only personnel trained and certified by NeuroQore will be permitted to administer treatment. All session and device information will be captured on appropriate data collection forms.

Study Duration:

The study is anticipated to last up to 6 months including enrollment and follow-up. Individual participant duration in the study will be 1 day of treatment, 24-hour and 7-day follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 22-85.
2. Current diagnosis of major depressive disorder according to the criteria defined in the current Diagnosis and Statistical Manual of Mental Disorders (DSM-V) without psychotic features.
3. Failed to receive satisfactory improvement from prior antidepressant medication in the current episode.
4. MADRS score > 20 at baseline and immediately prior to the day of treatment.
5. Agrees to adhere to the study treatment and follow-up schedule.
6. Willingness to remain on stable medications during rTMS therapy.
7. Fluent in English.

Exclusion Criteria:

1. Any medical conditions that would preclude the use of rTMS to treat depression.
2. Any conditions that would prevent the ability to undergo MRI testing.
3. Pregnancy as determined by serum/urine pregnancy test
4. History of epilepsy, seizure(s), or a seizure disorder as determined by the principal investigator based on a medical history obtained from the patient and/or others authorized to provide such history, combined with a brief screening instrument.
5. Active substance abuse
6. Diagnosis of bipolar or psychotic disorder
7. Considered to be at moderate-high risk of suicide according to the CSSRS assessment (i.e., Answers YES to Question 3 and NO to Question 6; or answers YES to Question 4, 5, or 6)
8. As determined by the Principal Investigator, subjects with cognitive impairment according to either the medical history obtained from the patient and/or a reliable secondary source, or the results of the Montreal Cognitive Assessment (MoCA) performed during screening.

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-01-16 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) Score | From enrollment to final MADRS score assessment within 2 weeks.
  Change in MADRS score from baseline to immediately post treatment, 24 hours and 7 days post-treatment

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) Score | From enrollment to final PHQ-9 score assessment within 2 weeks.
  Change in PHQ-9 score from baseline to immediately post treatment, 24 hours and 7 days post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- LGTC Group, San Jose, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
PII and Proprietary data will likely not be shared.